CLINICAL TRIAL: NCT02099045
Title: Initial Patient Evaluation in the Emergency Department With Point-of-Care Ultrasonography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Weile, MD, PhD student, Aarhus University Hospital
Other Study IDs: DNVK1305018
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Point of Care Ultrasonography in the Emergency Department.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ultrasound examination: All patients over the age of 18 presenting in the emergency department.
  Interventions: Device: Point of Care Ultrasonography

INTERVENTIONS:
Device: Point of Care Ultrasonography

SUMMARY:
Background: It is well known that emergency physicians can conduct ultrasound examinations as a supplement to initial physical examination. No previous studies have been conducted to evaluate the total findings with ultrasound on a broad unselected group of patients in the Emergency Department.

Aim: We aim to identify the pathology found in an unselected cohort of patients in a Rural Emergency Department. Secondarily we aim to quantify the changes done in treatment as a result of the ultrasound examination performed bedside in the Emergency Department.

Hypothesis: Supplemental ultrasonographical examination will change diagnostics and treatment in 10 % of an unselected cohort of patients in the Emergency Department.

Method: We will perform a structured ultrasound examination of 406 patients on an unselected cohort in the emergency department. All patients age 18 years and above presenting in the emergency department will be included in the study. Patients unwilling to give informed consent will be excluded from the study. Patients will be excluded if the ultrasonographic examination cannot be performed within the first two hours after initial contact with the treating physician. The study will be conducted in two substudies. Sub study 1 including all patient legally competent to give informed consent. Sub study 2 including all legally incompetent patients who cannot give informed consent due to acute illness. These patients will be included in the study under the rules of emergency research.

After including the patients we will ask the treating physician a series of binary questions regarding diagnosis and treatment plan.

Outcome: Primary outcome is the pathology found by ultrasound in the department. Secondary outcome will be the changes in diagnosis or treatment plan. Pathology and changes in diagnosis/treatment will be stratified according to initial complaint, triage level, age and other factors. This has never been done on unselected patients in the Emergency Department.

Ethical considerations and adverse effects: Ultrasound transmits high frequency waves into the tissue, which is reflected to the ultrasound probe. The time and magnitude of the returning sound waves are interpreted into picture on the screen. No adverse effects have been reported on the basis of the sound waves transmitted through the tissue.

Some patients might experience discomfort due to the sticky sensation from the application of ultrasound gel. Others might experience discomfort from the pressure applied to the probe under the imaging. Adverse effects, which we are not aware of, may exist. However, clinical ultrasound has existed since the 1950'ies and new adverse effects are unlikely.

Publication: All results will be published in international peer-review journals. Also in the event of inconclusive results.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 presenting at the ED

Exclusion Criteria:

* Sonographic examination cannot be performed within the first two hours
* Failure to consent.
* Sonographical examination interferes with lifesaving treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Unselected consecutive patients in the Emergency Department.
Sampling Method: Probability Sample
Enrollment: 406 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Pathology found by POC ultrasonography | Within two hours after initial evaluation of the patient.
  Cardiac function. Pericardial effusion more than 3 mm. Left ventricular function: Hyper dynamic, Normal, Mildly reduced, Moderately reduced, Severely reduced. Hypertrophic left ventricle: Ventricle wall > 1,2 cm Right ventricle function: TAPSE: > 20 mm: 16-20 mm: 13-15 mm: 10-12 mm: < 10 mm. Right ventricle wall > 0,8mm Left ventricle < right ventricle. Aortic sclerosis, Visible mass in lumen, Visible papillary muscle rupture, Pathology to mitral or tricuspid valve, Other findings. Inferior Vena Cava. IVC diameter : < 10 mm,10 -15mm, 16- 20mm, > 20mm IVC respiratory variation: collapse, > 50%, <50%, none Lung ultrasound: Absence of lung sliding, Visible pleural effusion, Multiple b-lines (≥3 in focal area) Abdominal ultrasound: Free fluid, Hydronephrosis: Left; Right, Gallbladder wall thickening > 4 mm Gallbladder width: > 4 cm,Murphey's sign, Visible cholecystolithiasis, Aortic aneurism: Size in cm Bladder size in ml Evaluation of the deep veins on the lower extremity for DVT

SECONDARY OUTCOMES:
Changes in diagnostics or treatments plan | Within 2 hours after primary evaluation of the patient after the ultrasound examination has been performed.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Bo Weile, MD, Principal Investigator — Research Center for Emergency Medicine; Hans Kirkegaard, MD, Professor, dr.med, ph.d., Study Chair — Research Center for Emergency Medicine; Erik Sloth, MD, professor, dr.med., ph.d, Study Chair — Department of Anaesthesiology, Skejby University Hospital; Christian Alcaraz Frederiksen, MD, PhD, Study Chair — Department of Cardiology, Aarhus University Hospital; Christian Laursen, MD, Study Chair — Department of Respiratory Medicine, Odense University Hospital
Locations (1):
- Emergency Department, Regional Hospital Herning, Herning, Denmark

REFERENCES:
- See also: Official site for Research Center for Emergency Medicine — http://akutforskning.au.dk/